CLINICAL TRIAL: NCT02369549
Title: Micro-Particle Curcumin for the Treatment of Chronic Kidney Disease
Acronym: MPAC-CKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Kidney Foundation of Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MPAC-CKD
Record Dates: First submitted 2015-01-13; First posted 2015-02-24 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease (CKD); Micro-particle curcumin; Albuminuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Albuminuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Micro-particle curcumin (Active Comparator): Three 30 mg capsules once daily, self-administered for 6 months.
  Curcumin is a nutraceutical, which are products isolated or purified from foods. The rhizomes of the plant Curcuma longa produces turmeric, a spice commonly used in Indian cuisine. Turmeric is comprised of three curcuminoids, of which curcumin is the most abundant. Curcumin is a polyphenol molecule that has been investigated for anti-inflammatory and anti-neoplastic properties since the 1970s.
  Interventions: Drug: Micro-particle Curcumin
- Placebo (Placebo Comparator): Three 30 mg capsules taken once daily, self-administered for 6 months.
  Placebo capsules are identical to the curcumin capsules in color, taste, smell, size and shape.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Micro-particle Curcumin — as described in Arm
  Other Names: Theracumin-Pro 300
  Arms: Micro-particle curcumin
Drug: Placebo — Looks, smells, tastes and feels exactly like the Curcumin capsules.
  Arms: Placebo

SUMMARY:
An investigator initiated pilot trial: two arm, double blind, placebo controlled, randomized, parallel group of approximately 750 patients with chronic kidney disease, and who have evidence of overt proteinuria, will be treated with micro-particle curcumin versus placebo over 24 weeks from start of the investigational medication date (approximately 6 months) to test whether curcumin can slow chronic kidney disease progression in patients. Three 30 mg capsules of micro-particle curcumin will be self-administered once daily in the morning to determine the the safety and efficacy of curcumin relative to placebo in reducing albuminuria and slowing the loss of eGFR.

DETAILED DESCRIPTION:
Limiting the progression from CKD to end-stage renal disease is one of the most important goals in kidney medicine. The evidence implicating inflammation and fibrosis in that process is strong, and there is abundant mechanistic and animal model data to show that curcumin is a potent inhibitor of both inflammation and fibrosis. Two preliminary randomized trials in human CKD hint at curcumin's enormous therapeutic potential in CKD. The Principal Investigator/Sponsor will rigorously test this potential in a broadly selected sample of up to 750 patients with CKD. Compared to previous studies, this study's results will be generalizable across other etiologies of CKD and with a larger sample size; this study will provide more precise estimates of curcumin's benefits and risks. Also, this study proposes to use a new, micro-particle formulation of curcumin that is highly bioavailable. The Principal Investigator/Sponsor will assess curcumin's effects on three key markers of kidney health that encompass the cardinal functions of the nephron. Positive results from MPAC-CKD will lay solid scientific ground-work for a multi-centre trial capable of testing micro-particle curcumin's effect of the most meaningful outcomes: death and the development of end-stage renal disease.

To ensure that this study will have the necessary adherence and tolerability data, up to 750 patients with proteinuric CKD will be randomly assigned to 90 mg per day of micro-particle curcumin or matching placebo, for a total of 24 weeks (approximately 6 months). In the last few years, new formulations of curcumin have been shown to substantially augment absorption by improving its aqueous solubility. The micro-particle formulation of curcumin is one of these new formulations and is the only curcumin delivery system proven to increase bioavailability. Compared to traditional curcumin, micro-particle curcumin achieves total serum concentrations that are 27 fold higher. In this study, micro-particle curcumin will allow the study team to administer the equivalent of 3000 mg of traditional curcumin (which would require six 500 mg capsules daily), in a single 90 mg capsule. In addition, as opposed to traditional curcumin, there is no requirement to take micro-particle curcumin on a full stomach. The Investigator/Sponsor has selected a dose equivalent to 3 grams per day of curcumin because this is within the range of doses proven safe and effective and it will minimize pill burden by allowing the full daily dose to be achieved by three small 30 mg capsules daily In rare cases, curcumin has been reported to cause minor nausea, headache, diarrhea, yellow stool, and temporary giddiness. All unexpected reactions reported in previous studies were easily managed and happened at higher doses than what will be used in MPAC-CKD.

This study will assess two primary outcomes: the 6-month change in albuminuria, and the 6-month change in eGFR.

Secondary outcomes will include health-related quality of life, glycemic control among patients with diabetes mellitus, and a composite of progressive CKD, ESRD and death. The investigators will also measure serum curcumin levels in the first 30 randomized participants, who will have a 4.5 ml blood sample taken at the 12 week (3 month) visit. This sample will be processed and stored at -80 degrees C. for batch testing for plasma micro-particle curcumin concentrations.

The investigators will conduct a subgroup analysis based on participants 2-year risk of requiring dialysis using the validated Kidney Failure Risk Equation to group patients into a high risk group (10% or greater risk of dialysis within 2 years) and low risk group (<10% risk within 2 years).

Medical history, lab values and vitals will be collected and/or updated at each in-person visit. Each participant will be provided with instructions and study schedule. Participants with diabetes mellitus will be given a home glucose log-book.

Protocol compliance will be tested through pill counts and interviews at each follow-up visit. Side effects will be assessed using standardized case report forms at each visit. Participants will be contacted by telephone one week into the trial and then once every 4 weeks (monthly) for 28 weeks (approximately 7 months) for safety monitoring and reporting and to reinforce importance of compliance. In-person visits will occur at 12 and 24 weeks (approximately 3 and 6 months) after randomization and the start of the investigational medication, at which time investigational medication will be counted and supply replenished. First morning at-home urine specimens will be collected at baseline and again arranged at the in-person visits at 12 and 24 weeks (approximately 3 and 6 months). Participants will also be encouraged to report any events they may experience directly to the coordinator(s) and/or PI.

Participants who withdraw consent to continue treatments, will be encouraged to undergo the planned assessments. Withdrawal at the request of investigators or medical personnel may include, but are not limited to:

1. Symptoms are deemed to be potentially related to the sue of the investigational medication;
2. New diagnosis of exclusion criteria;
3. Inter-current illness not related to the use of the investigational Natural Health Product (NHP) medication;
4. Unacceptable side effects;
5. Death;
6. Improved health status.

Estimated time to complete recruitment: Averaging 136 weeks, approximately 34 months.

Long-term outcomes will be tracked using administrative data housed at The Institute for Clinical Evaluative Sciences (ICES), an independent research facility in Toronto, Ontario. ICES works with the Ontario Ministry of Health and Long-Term Care to study the impact of health care and diseases in Ontario.

A panel of external experts and study investigators will comprise the Steering Committee and will ensure the integrity of the study. They will be responsible for reviewing and acting upon the recommendations of the Data Safety Monitoring Board, amendments to the protocol, oversight of publication and dissemination of study results.

ELIGIBILITY:
Inclusion Criteria:

1. eGFR between 15 and 60 ml/min/1.73 m2;
2. Albuminuria, defined by the most recent measurement within the prior 3 months showing either: a) 24-hour urine collection with a minimum of 300 mg of protein, OR b) urinary albumin to creatinine ratio equivalent to a daily excretion of albumin of at least 300 mg;
3. If diabetic, is able and willing to take and record glucose levels at home;
4. If receiving and ACE inhibitor or angiotension II receptor blocker (ARB), the dosage must be stable for 2 weeks prior to screening. Patients not taking and ACE or ARB must have a documented medical contraindication (e.g. hyperkalemia, hypotension);
5. Willing and able to give written informed consent for participation and provide consent for access to medical data according to local data protection laws and regulations.

Exclusion Criteria:

1. Life expectancy < 1 year;
2. Known allergy to turmeric or its derivatives (ginger, curry, cumin, or cardamom);
3. Known allergy to ingredients of the study product or placebo (microcrystalline cellulose, vegetarian capsule, vegetable grade magnesium stearate, silica;
4. Pregnant or breastfeeding;
5. Women of child-bearing potential who are not either surgically sterile or not postmenopausal for at least 1 year;
6. Plans for transplantation during the study period;
7. Receipt of hemodialysis or peritoneal dialysis in the past 3 months;
8. Active peptic ulcer disease;
9. Hepatobiliary disease in the past 4 weeks;
10. Evidence of acute kidney injury (>50% increase in serum creatinine in the past 30 days);
11. History of significant bleeding (GI or retroperitoneal bleed requiring transfusion, or any intracranial hemorrhage in the past 6 months);
12. Ongoing use of warfarin;
13. Ongoing treatment with cyclophosphamide, camptothecin, mechlorethamine or doxorubicin;
14. Ongoing use of anti-psychotic medication including haloperidol, aripiprazole, risperidone, ziprasidone, pimozide, and quetiapine;
15. Previous participation in MPAC-CKD;
16. Current participation on another investigational medication trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Change in albuminuria from baseline to 24 week (6 month) | Baseline and 24 weeks (6 months)
  Albuminuria will be measured using urinary albumin-to-creatinine ratio from first morning urine samples. At each visit (pre-randomization, and 3- and 6-months post-randomization), urinary albumin-to-creatinine ratio is measured on two consecutive days and the average of the two values will be computed. The average of the two values will be log-transformed using the natural logarithm. Albuminuria is the cardinal manifestation of a malfunctioning filtration barrier and the spillage of albumin into renal tubules is thought to be toxic to tubular cells, resulting in further kidney damage. Therefore, in the current understanding, albuminuria is both a marker and a mediator of kidney damage. Reduction of albuminuria has repeatedly been associated with improved renal outcomes. Leaders in the field of nephrology recommend that albuminuria be used as a valuable predictor of response to therapy for the prevention of kidney failure.
Change in Estimated Glomerular Filtration rate (eGFR) from baseline to 24 weeks (6 months) | Baseline and 24 weeks (6 months)
  eGFR will be calculated using the CKD-EPI formula. The investigators will estimate the between-group difference in change in eGFR (6-month eGFR minus baseline eGFR), expressed in mL/min per 1.73m2, using linear regression.

SECONDARY OUTCOMES:
Change in glycemic control among participants with diabetes mellitus | Baseline and 24 week (6 months)
  The investigators will summarize the percentage of glycated hemoglobin pre-randomization and 6-months post-randomization and will present the between-group difference in change in percentage of glycated hemoglobin (6-month value minus pre-randomization value) among patients with diabetes mellitus.
Renal failure composite | 24 week (6 months)
  The investigators will report on the outcome of progressive CKD, ESRD, and death, first as a composite outcome, and then as separate components. ESRD will be defined as an eGFR <15 mL/min/1.73 m2 or the initiation of renal replacement therapy, which includes chronic dialysis or transplantation; progressive CKD will be defined as an eGFR loss of ≥ 30% (anytime during follow-up from the pre-randomization baseline value) or ESRD. Less than 10% of participants will be expected to experience these outcomes by 6 months. The focus of this analysis is to document any trends to inform the expected event rate for future studies.
Change in health-related quality of life (physical composite summary) | Baseline and 24 week (6 months)
  Health-related quality of life scores will be determined by the RAND version of the 36-Item Short Form Health Survey (SF-36) administered pre-randomization and at 3-months and 6-months post-randomization. The physical composite summary (PCS) score of the SF-36 will be examined. The between-group difference in change in score, 6-month value minus pre-randomization value, will be reported with 95% CIs.
Change in health-related quality of life (mental composite summary) | Baseline and 24 week (6 months)
  Health-related quality of life scores will be determined by the RAND version of the 36-Item Short Form Health Survey (SF-36) administered pre-randomization and at 3-months and 6-months post-randomization. The mental composite summary (MCS) score of the SF-36 will be examined. The between-group difference in change in score, 6-month value minus pre-randomization value, will be reported with 95% CIs.

OTHER OUTCOMES:
Serum curcumin levels | 12 weeks (3 months)
  To confirm our micro-particle curcumin was bioavailable, and to strengthen any relationship between micro-particle curcumin and any outcomes identified, serum levels of curcumin and its major metabolites will be measured in the first 30 participants 3 months after randomization (including patients taking micro-particle curcumin and those taking placebo). Serum curcumin and its major metabolites will be summarized in the first 30 participants randomized, by group. The between-group difference in average serum curcumin levels measured 3-months post-randomization will be reported with the 95% CI.
Kidney failure risk subgroup | Baseline and 24 week (6 months)
  The investigators will conduct an exploratory subgroup analysis based on a higher or lower estimated risk of kidney failure, using the kidney failure risk equation. Participants with a 2-year risk of ESRD less than 10% will be classified as lower risk, and patients with a risk of 10% or more will be classified as higher risk.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Weir, Nephrologist, Principal Investigator — LHSC
Locations (4):
- Canada (4):
  - Population Health Research Institute, Hamilton, Ontario
  - Kidney Clinical Care Unit, London, Ontario
  - University Hospital, London, Ontario
  - Victoria Hospital, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weir MA, Walsh M, Cuerden MS, Sontrop JM, Urquhart BL, Lim YJ, Chambers LC, Garg AX. The effect of micro-particle curcumin on chronic kidney disease progression: the MPAC-CKD randomized clinical trial. Nephrol Dial Transplant. 2023 Sep 29;38(10):2192-2200. doi: 10.1093/ndt/gfad037. PMID 36849161
- [Derived] Weir MA, Walsh M, Cuerden MS, Sontrop JM, Chambers LC, Garg AX. Micro-Particle Curcumin for the Treatment of Chronic Kidney Disease-1: Study Protocol for a Multicenter Clinical Trial. Can J Kidney Health Dis. 2018 Dec 5;5:2054358118813088. doi: 10.1177/2054358118813088. eCollection 2018. PMID 30619615

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT02369549/Prot_SAP_000.pdf